CLINICAL TRIAL: NCT01886937
Title: The Quantification of Ingestive Behavior
Brief Title: Studying the Effects of Phentermine on Eating Behavior
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 6415
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Phentermine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 37.5 mg Phentermine daily for 7 days (Experimental): In this arm, participants receive 37.5mg phentermine for one week followed by 2 weeks of placebo.
  Other names for phentermine:
  adipex ionamin
  Interventions: Drug: Phentermine
- Placebo (for phentermine 37.5mg) (Placebo Comparator): In this arm, participants receive Placebo (for 37.5mg phentermine) for two weeks followed by phentermine 37.5mg for 7 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Phentermine — After 7 days of phentermine 37.5 mg administration, food intake should be less than after 14 days of placebo.
  Other Names: adipex; ionamin
  Arms: 37.5 mg Phentermine daily for 7 days
Drug: placebo — Food intake as measured by a laboratory study should be greater after 7 days of placebo administration compared to seven days of phentermine administration.
  Other Names: sugar pill
  Arms: Placebo (for phentermine 37.5mg)

SUMMARY:
The goal of this study is to determine whether one week of phentermine compared to placebo administration results in changes in food intake during a laboratory meal.

DETAILED DESCRIPTION:
This study aims to explore whether short-term measures of eating behavior can be related to later, longer-term weight loss. In a double-blind, randomized fashion, participants will be asked to take study medication for three weeks: one week of phentermine and two weeks of placebo. At the end of the first and third weeks, participants will be asked to participate in a range of eating behavior studies. Following this three-week, double-blind phase, participants will be offered 6 months of open treatment for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-40kg/m2
* Stable weight (+5 lbs) for a minimum of 3 months
* Systolic Blood Pressure <140mm Hg
* Diastolic Blood Pressure <90 mm Hg
* Pulse <95 beats per minute
* English language proficiency

Exclusion Criteria:

* Previous unsuccessful trial of phentermine
* Prior adverse reaction to phentermine
* On any antidepressant medications,especially monoamine oxidase inhibitors(MAOI)
* History of neurological disorder (e.g. dementia)
* History of moderate or severe head injury
* Current or past history of coronary artery disease
* Current or past history of stroke or transient ischemic attack
* Current or past history of heart arrhythmias
* Current of past history of congestive heart failure
* Current or past history of peripheral artery disease
* Current or past history of liver disease
* Current or past history of kidney disease
* Uncontrolled diabetes mellitus (type I or II)
* Narrow-angle glaucoma
* Hypo- or hyper-thyroidism not adequately treated
* On medications (prescribed or OTC) known to affect appetite (e.g. diet pills), weight, or metabolism
* Current or past history (within the past 12 months) of major depression
* Current or past history (past 12 months) of alcohol or drug abuse or dependence
* Current or past history (lifetime) of amphetamine abuse or dependence
* Known history of learning disorder or developmental disability
* Current or past Attention Deficit Hyperactivity Disorder (ADHD)
* Pregnancy, planning to become pregnant, or lactation within the previous 6 months
* Waist circumference greater than 188cm
* Indwelling metallic object (e.g., pacemaker,pump), non-removable metal jewelry, medicinal patch or recent metallic ink tattoo
* Significant claustrophobia
* Current or past history of anorexia nervosa,bulimia nervosa (within the past 12 months) or binge eating disorder (within the previous 6 months)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Mayer, MD, Principal Investigator — Columbia University Medical Center/New York State Psychiatric Institute
Locations (1):
- The New York State Psychiatric Institute at Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 patients were screened for eligibility between July 2012 and July 2013 at an academic medical center in New York City, NY.
Pre-assignment Details: 13 of the 37 participants were randomized. Of those not randomized, 18 did not meet inclusion criteria and 6 chose not to participate.
Groups:
- 37.5 mg Phentermine Daily for 7 Days First,Followed by Placebo: In this arm, participants receive 37.5mg phentermine for one week followed by 2 weeks of placebo.
  Other names for phentermine:
  adipex ionamin
  Phentermine: After 7 days of phentermine 37.5 mg administration, food intake should be less than after 14 days of placebo.
- Placebo (for Phentermine 37.5mg) First, Followed by Phentermin: In this arm, participants receive Placebo (for 37.5mg phentermine) for two weeks followed by phentermine 37.5mg for 7 days.
  placebo: Food intake as measured by a laboratory study should be greater after 7 days of placebo administration compared to seven days of phentermine administration.
Period: Overall Study
Arm/Group | 37.5 mg Phentermine Daily for 7 Days First,Followed by Placebo | Placebo (for Phentermine 37.5mg) First, Followed by Phentermin
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 37.5 mg Phentermine First, Then Placebo: In this arm, participants receive 37.5mg phentermine for one week followed by 2 weeks of placebo.
  Other names for phentermine:
  adipex ionamin
  Phentermine: After 7 days of phentermine 37.5 mg administration, food intake should be less than after 14 days of placebo.
- Placebo First, Then 37.5mg Phentermine: In this arm, participants receive Placebo (for 37.5mg phentermine) for two weeks followed by phentermine 37.5mg for 7 days.
  placebo: Food intake as measured by a laboratory study should be greater after 7 days of placebo administration compared to seven days of phentermine administration.
- Total: Total of all reporting groups
Arm/Group | 37.5 mg Phentermine First, Then Placebo | Placebo First, Then 37.5mg Phentermine | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14) | 37 (16) | 42 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 0

OUTCOME MEASURES:

1. Primary Outcome: Food Intake
Description: The primary outcome measure is food intake assessed by laboratory meal study after one week of phentermine administration compared to one week of placebo administration.
Time Frame: one week
Population: This is a cross over design study. All participants received phentermine and placebo.The phentermine arm listed here includes all participants who received phentermine (regardless of whether they received it first or second). The placebo arm includes all those who received placebo (regardless of whether they received placebo first or second).
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- 37.5 mg Phentermine Daily for 7 Days: In this arm, participants receive 37.5mg phentermine for one week .
  Other names for phentermine:
  adipex ionamin
  Phentermine: After 7 days of phentermine 37.5 mg administration, food intake should be less than after 14 days of placebo.
- Placebo (for Phentermine 37.5mg): In this arm, participants receive Placebo (for 37.5mg phentermine) for 7 days.
  placebo: Food intake as measured by a laboratory study should be greater after 7 days of placebo administration compared to seven days of phentermine administration.
Arm/Group | 37.5 mg Phentermine Daily for 7 Days | Placebo (for Phentermine 37.5mg)
Number analyzed (Participants) | 13 | 13
kcal | 849 (572) | 975 (504)
Statistical Analysis 1: Comparison: 37.5 mg Phentermine Daily for 7 Days vs Placebo (for Phentermine 37.5mg); Test type: Superiority; p = 0.26, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: One week for each study intervention (phentermine or placebo).
Groups:
- 37.5 mg Phentermine: This describes all participants who received 37.5mg phentermine for one week.
  Other names for phentermine:
  adipex ionamin
- Placebo: This group refers to all participants who received Placebo.
Arm/Group | 37.5 mg Phentermine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 9/13 | 8/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 37.5 mg Phentermine (N=13) | Placebo (N=13)
headache (Nervous system disorders) | 2 | 3
constipation (Gastrointestinal disorders) | 3 | 4
nausea (Gastrointestinal disorders) | 2 | 1
feeling drowsy or sleepy (Nervous system disorders) | 1 | 1
increased appetite (Gastrointestinal disorders) | 0 | 2
trouble concentrating (Nervous system disorders) | 2 | 1
irregular heartbeat (Cardiac disorders) | 0 | 1
diarrhea (Gastrointestinal disorders) | 0 | 1
dry mouth (General disorders) | 5 | 3
decreased appetite (Gastrointestinal disorders) | 5 | 3
tremor (Nervous system disorders) | 2 | 1
dizziness (Nervous system disorders) | 2 | 1
lightheaded upon standing (Nervous system disorders) | 2 | 1
difficulty sleeping (Nervous system disorders) | 3 | 4
sour taste (Gastrointestinal disorders) | 1 | 0
increased urination (Renal and urinary disorders) | 2 | 3
shortness of breath (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No